CLINICAL TRIAL: NCT01815632
Title: Assessment of Bone Marrow-derived Cellular Therapy in Progressive Multiple Sclerosis (ACTiMuS)
Acronym: ACTiMuS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Bristol NHS Trust (Other)
Collaborators: Bristol Royal Hospital for Children (Other); University of Bristol (Other); University of Nottingham (Other); NHS Blood and Transplant (Other Government); Kenneth and Claudia Silverman Family Foundation (Other); Multiple Sclerosis Trust (Unknown); Medical Research Council (Other Government); Rosetrees Trust (Other); Catholic Bishops of England and Wales (Unknown); Friends of Frenchay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTiMuS; ISRCTN27232902 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Progressive Multiple Sclerosis
Keywords: multiple sclerosis; progressive MS; stem cell; cell therapy; neurodegeneration; CNS repair
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early infusion of autologous marrow (Experimental): Intravenous infusion of autologous bone marrow (without myeloablation) on the day of bone marrow harvest. Infusion of autologous blood at one year post-harvest
  Interventions: Other: Early infusion of autologous marrow
- Late infusion of autologous marrow (Experimental): Intravenous infusion of autologous blood on the day of bone marrow harvest. Infusion of autologous bone marrow (without myeloablation) at one year post-harvest
  Interventions: Other: Late infusion of autologous marrow

INTERVENTIONS:
Other: Early infusion of autologous marrow — Intravenous infusion of autologous bone marrow without prior myeloablation on the day of bone marrow harvest and infusion of autologous blood at one year post-bone marrow harvest
  Arms: Early infusion of autologous marrow
Other: Late infusion of autologous marrow — Infusion of blood on day of bone marrow harvest with intravenous infusion of autologous bone marrow without prior myeloablation one year post-bone marrow harvest.
  Arms: Late infusion of autologous marrow

SUMMARY:
Multiple sclerosis - MS - affects 1.3m people worldwide, costing the European Union economy €9 billion/year, through both direct and indirect consequences of progressive disability. Despite the usual relapsing-remitting presentation, over 80% of patients develop progressive disability; 40% require a wheelchair within 10 years of diagnosis. At present, there are no treatments that reverse, halt or even slow progressive disability in MS.

The investigators recently completed one of the first feasibility/safety trials in the world of reparative bone marrow cell therapy in 6 patients with longstanding MS (www.nature.com/clpt/journal/v87/n6/full/clpt201044a.html). Safety was confirmed, and intensive repeated tests on the patients measuring nerve conduction in various pathways in the brain and in the spinal cord showed statistically significant improvements at 12 months in every patient. While highly preliminary and involving only a very small number of patients, these results at least raise the possibility of a significant (though very partial) underlying repair effect within the damaged nervous system.

The investigators believe this urgently requires further testing - both to accelerate benefit for patients, and to begin improving therapeutic efficacy. The investigators therefore propose a programme of translational and clinical stem cell research, aiming (1) to continue translation with a phase two controlled trial of bone marrow cells in patients with longstanding MS; and (2) to explore in parallel the potential mechanisms of action, by studying bone marrow cells from treated patients and control subjects, aiming to establish which of the various relevant bone marrow subpopulations contribute to efficacy, and which particular reparative mechanism(s) are important. The investigators hope these studies will not only confirm the therapeutic benefit of this approach, but also provide the basis for improving the magnitude and impact of this novel and exciting treatment modality.

DETAILED DESCRIPTION:
The primary objective is to determine whether autologous bone marrow (BM) (ie taken from the patients themselves rather than from a BM donor) cell therapy is truly beneficial in chronic multiple sclerosis - as our small, uncontrolled phase 1 trial suggested (www.nature.com/clpt/journal/v87/n6/full/clpt201044a.html).

The investigators also aim to answer the following questions:

1. Do BM mesenchymal stem cells from patients with MS differ in the range or extent of reparative and neuroprotective properties from those from control individuals?
2. What reparative and neuroprotective properties do BM stem cell subpopulations other than mesenchymal stem cells possess, and do these differ between MS patients and controls?
3. Can BM stem cell subpopulations be isolated from blood samples from MS patients following treatment, and, if so, for how long?

Bone marrow contains stem cells capable of replacing all the cells in the blood. Recently, bone marrow has been found to contain cells capable of replacing cells in tissues and organs other than blood. In addition, infusion of bone marrow-derived cells has been shown to have significant effects on the immune system and to promote the survival of central nervous system cells under toxic conditions. These properties are of considerable interest to those working to develop cell-based therapies for neurodegenerative disease.

The potential of such cells to aid repair in multiple sclerosis (MS) has been examined in experimental models of MS. Myelin is the substance that insulates neurons within the central nervous system and is attacked in MS. Infusion of adult bone marrow cells into a vein aids myelin repair (remyelination) in these models of MS. Recently, the investigators performed a small pilot study to examine the effects of harvesting bone marrow from MS patients and infusing this back into each patient's vein. This was well tolerated and no significant adverse events were encountered. Electrophysiological studies appeared to show some improvement but, given the small numbers of participants in the phase 1 trial, no definitive conclusion can be made regarding this.

The current study seeks to address the question of whether genuine improvements in neurophysiological tests are seen in MS patients with progressive disease following infusion of bone marrow.

A prospective, randomised, double-blind, placebo-controlled, stepped wedge design will be employed at a single centre (Bristol, UK). Eighty patients with progressive MS will be recruited; 60 will have secondary progressive disease (SPMS) but a subset (n=20) will have primary progressive disease (PPMS). Participants will be randomised to either early (immediate) or late (1 year) intravenous infusion of autologous, unfractionated bone marrow. The placebo intervention is infusion of autologous blood. The primary outcome measure is global evoked potential derived from multimodal evoked potentials. Secondary outcome measures include adverse event reporting, clinical (EDSS and MSFC) and self-assessment (MSIS-29) rating scales, optical coherence tomography (OCT) as well as brain and spine MRI. Participants will be followed up for a further year following the final intervention. Outcomes will be analyzed on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically-definite MS as defined by the McDonald criteria
* Aged 18 - 65 years.
* EDSS of 4.0 to 6 inclusive
* Disease duration >5 years
* Disease progression (increase in physical disability, not due to major relapse) in preceding year
* Signed, written informed consent
* Willing and able to comply with study visits according to protocol for the full study period

Exclusion Criteria:

* Pregnancy, breastfeeding or lactation
* History of autologous/allogenic bone marrow transplantation or peripheral blood stem cell transplant
* Bone marrow insufficiency
* History of lymphoproliferative disease or previous total lymphoid irradiation
* Immune deficiency
* Current or recent (<5 years) malignancy
* Chronic or frequent drug-resistant bacterial infections or presence of active infection requiring antimicrobial treatment
* Frequent and/or serious viral infection
* Systemic or invasive fungal disease within 2 years of entry to study
* Significant renal, hepatic, cardiac or respiratory dysfunction
* Contraindication to anaesthesia
* Bleeding or clotting diathesis
* Current or recent (within preceding 12 months) immunomodulatory therapy other than corticosteroid therapy
* Treatment with corticosteroids within the preceding three months
* Significant relapse within preceding 6 months
* Predominantly relapsing-remitting disease over preceding 12 months
* Radiation exposure in the past year other than chest / dental x-rays
* Previous claustrophobia
* The presence of any implanted metal or other contraindication to MRI
* Participation in another experimental study or treatment within the preceding 24 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Global evoked potential (GEP): mean change from time of marrow infusion to end of study | Entry and every 6 months for 2 years
  Multimodal evoked potentials will be examined at 0, 6, 12, 18 and 24 months. Evoked potential abnormalities will be quantified according to a 4-point graded ordinal score modified from Leocani et al (JNNP 2006, 77:1030-1035) (0=normal; 1=increased latency; 2=increased latency and abnormal amplitude; 3=absent).
  The recording of the evoked potentials shall be in accordance with the Guidelines of the International Federation of Clinical Neurophysiology and analysis will be performed using standard methods. Electrophysiological responses shall be considered abnormal if they exceed 2.5 standard deviations of the normal values or cannot be detected.

SECONDARY OUTCOMES:
Safety | Continuous throughout study period (2 years)
  Evaluation of number and nature of adverse events
Expanded disability status scale | At entry then 6 weeks, 6 months and 1 year after each infusion
  Time to EDSS progression of at least one point from a baseline EDSS of 4.0, 4.5 or 5.0 or at least 0.5 points from a baseline EDSS ≥5.5
Multiple sclerosis impact scale (MSIS-29) | At entry then 6 weeks, 6 months and 1 year after each infusion
  Mean change from baseline to end of study on the patient-based MSIS-29 scale
Multiple sclerosis functional composite (MSFC) | At entry then 6 weeks, 6 months and 1 year after each infusion
  Mean change on MSFC score from baseline to final visit
MRI head and cord | At entry, 1 year and 2 years post-harvest
  The secondary MRI outcome measures will relate to 1) lesion load, 2) atrophy measures both of the brain and of cross-sectional area of the spinal cord, and changes in mean diffusivity.
  Exploratory analysis of the resting-state fMRI data will investigate correlations between network patterns and 'strength' of networks connectivity from the resting-state fMRI with classifications revealed by the various evoked potential studies
Optical coherence tomography | Entry, 1 year and 2 years post-harvest
  Measurement of retinal nerve fibre layer thickness and macular volume

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Scolding, FRCP PhD, Principal Investigator — University of Bristol & North Bristol NHS Trust
Locations (1):
- Southmead Hospital, Bristol, United Kingdom

REFERENCES:
- [Derived] Rice CM, Marks DI, Ben-Shlomo Y, Evangelou N, Morgan PS, Metcalfe C, Walsh P, Kane NM, Guttridge MG, Miflin G, Blackmore S, Sarkar P, Redondo J, Owen D, Cottrell DA, Wilkins A, Scolding NJ. Assessment of bone marrow-derived Cellular Therapy in progressive Multiple Sclerosis (ACTiMuS): study protocol for a randomised controlled trial. Trials. 2015 Oct 14;16:463. doi: 10.1186/s13063-015-0953-1. PMID 26467901